CLINICAL TRIAL: NCT01666717
Title: Characterization of Disease Related Changes in Inflammatory Bowel Disease Using Fecal Metabolite Profiling
Status: Completed | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Kristin Verbeke, Professor K. Verbeke, KU Leuven
Other Study IDs: ML4355_VOC
Record Dates: First submitted 2012-08-14; First posted 2012-08-16 (Estimated); Last update posted 2012-08-17 (Estimated); Status verified 2012-08

CONDITIONS: Inflammatory Bowel Diseases
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Fecal samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Healthy controls (HC): HC
- Inflammatory Bowel Disease (IBD) patients: Crohn's disease (CD), Ulcerative colitis (UC) and pouchitis

SUMMARY:
The purpose of the study is to evaluate fecal metabolites profiles of Inflammatory Bowel Disease(IBD) patients versus healthy controls (HC).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of IBD
* Age >18 years

Exclusion Criteria:

* Use of antibiotics in the preceding month
* Intake of pre- or probiotics

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Primary care clinic
Sampling Method: Probability Sample
Enrollment: 204 (Actual)
Dates: Start 2008-08; Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- KULeuven-UZLeuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] De Preter V, Machiels K, Joossens M, Arijs I, Matthys C, Vermeire S, Rutgeerts P, Verbeke K. Faecal metabolite profiling identifies medium-chain fatty acids as discriminating compounds in IBD. Gut. 2015 Mar;64(3):447-58. doi: 10.1136/gutjnl-2013-306423. Epub 2014 May 8. PMID 24811995